CLINICAL TRIAL: NCT05386459
Title: Prospective Two-week Open-label Application Experimental Randomized Single-center Non-interventional Study of the Drug Ingaron in Patients With a New Coronavirus Infection COVID-19
Brief Title: Study of the Use of the Drug Ingaron in Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: SPP Pharmaclon Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2GAMMACOVID-19
Record Dates: First submitted 2022-05-20; First posted 2022-05-23 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: COVID-19 Respiratory Infection; Viral Pneumonia
Keywords: COVID-19 treatment; interferon gamma
MeSH Terms: conditions — Pneumonia, Viral | interventions — Interferon-gamma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Main: Ingaron (INN: recombinant human interferon gamma, lyophilizate for solution preparation for intramuscular and subcutaneous administration 500,000 IU) 1 subcutaneous injection 1 time per day (in the morning) daily for 5 days (5 injections in total) against the background of basic antibacterial and symptomatic therapy
  Interventions: Drug: Interferon Gamma
- Control: Only basic antibacterial and symptomatic therapy. The use of the study drug was carried out on the basis of the decision of the medical commission with the execution of the protocol and primary medical documentation of the patient

INTERVENTIONS:
Drug: Interferon Gamma — injection form
  Other Names: Ingaron; Interferon gamma human recombinant
  Groups: Main

SUMMARY:
Interferon gamma is a powerful endogenous regulatory cytokine that activates the antiviral immune response, while it also has its own antiviral activity. The objective of this study was to evaluate the effectiveness of the proposed treatment regimen with Ingaron (INN: recombinant interferon gamma human, lyophilisate for preparing a solution for intramuscular and subcutaneous administration of 500,000 IU) in patients with viral pneumonia.

DETAILED DESCRIPTION:
The study drug was prescribed for therapeutic purposes according to the following scheme:

500,000 IU s / c 1 time per day daily for 5 days. A total of 4 visits were scheduled. Visits 0 and 1 could be combined provided that the chronological sequence of screening and randomization procedures was followed.

The main stages of the study:

screening - lasting no more than 1 day; treatment - within 10-14 days, including the use of the investigational medicinal product for 5 days (from the first day of the basic therapy, daily).

The total duration of observation is up to 14 days. Patients who completed participation in the study or dropped out of the study ahead of schedule were followed up by the attending physician in accordance with the rules for managing such patients for a medical institution.

ELIGIBILITY:
Inclusion Criteria:

* Patients with viral pneumonia according to CT scan, regardless of:

  * degree of damage to the lungs;
  * results of a laboratory test for the presence of SARS-CoV-2 RNA;
  * epidemiological history.
* Patients of both sexes over 18 years of age.
* Patients who are able to read, understand and independently certify in writing the informed consent form.
* Negative pregnancy test for female patients of reproductive age with preserved reproductive function.

Exclusion Criteria:

* Any clinically confirmed or documented history of disease that may make it difficult to interpret the data being assessed.
* No symptoms of a respiratory infection.
* Severe liver or kidney failure, and/or failure of other vital organs, in the stage of decompensation (kidney - creatinine level> 2X ULN, liver tests: liver enzymes (AST and ALT) > 3X ULN).
* Diseases of the central nervous system with severe impairment of intellectual and mnestic functions.
* Any other disease or condition that, in the opinion of the investigator, may confound the results of the study, limit the patient's participation in the study, or place the patient at greater risk.
* Serious diseases and pathological conditions (PE, oncological diseases, etc.) that require emergency medical care or threaten the patient's life.
* Mild, subclinical, asymptomatic or severe form of the course of the disease.
* Acute respiratory distress syndrome, sepsis, septic shock.
* Contraindications to the use of the investigational medicinal product.
* Individual intolerance to the ingredients that make up the study drug.
* Participation in any clinical trial within 1 month prior to baseline visit (Day 0-1).
* Pregnancy or breastfeeding.

Ages: 38 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with novel coronavirus infection COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Comparative analysis between treatment groups on the WHO Clinical Improvement Scale | Day 14
  The assessment was carried out according to the WHO Clinical Improvement Scale from 0 points - not infected, no manifestations or virological signs of infection, up to 8 points - died, death

SECONDARY OUTCOMES:
Difference between laboratory LDH values | Day 14
  Difference between laboratory LDH values compared to baseline
Difference between laboratory CRP values | Day 14
  Difference between laboratory CRP values compared to baseline
Difference between laboratory ferritin values | Day 14
  Difference between laboratory ferritin values compared to baseline
Changes in laboratory parameter D-dimer | Day 14
  Changes in laboratory parameter D-dimer compared with baseline
Comparative analysis of survival between treatment groups | Day 14
  Comparative assessment of CFR mortality rates
Comparative analysis of survival between treatment groups | Day 14
  Comparative assessment of IFR mortality rates
Change from baseline patient ratings of subjective outcomes based on various measures | Day 14
  Change from Baseline Patients in Subjective Outcomes Based on: Pulse Oxygen Saturation
Change from baseline patient ratings of subjective outcomes based on various measures | Day 14
  Change from baseline patient assessments of subjective outcomes based on the indicator: body temperature
Change from baseline patient ratings of subjective outcomes based on various measures | Day 14
  Change from Baseline Patients in Subjective Outcomes Based on Indicator: Blood Pressure
Comparative analysis between groups by indicators | Day 14
  Comparative analysis between groups by indicators: duration of fever
Comparative analysis between groups by indicators | Day 14
  Comparative analysis between groups by indicators: duration of hospitalization
Comparative analysis between groups on NEWS-2 indicators | Day 14
  Comparative assessment of the score according to the National Early Warning Rating 2 (NEWS-2), where the minimum score is 0, which corresponds to the general rules for managing a patient, from 7 points or more - emergency medical care is required in the ICU
Comparative analysis of the incidence and severity of adverse events | Day 14
  Comparative analysis of the incidence and severity of adverse events according to CTCAE version 4.03 of 2010

CONTACTS AND LOCATIONS:
Overall Officials: Anatoly I Saulin, Master, Study Director — SPP Pharmaclon Ltd.
Locations (1):
- City Clinical Hospital named after M.E. Zhadkevich Moscow City Health Department, Moscow, Russia

REFERENCES:
- [Result] Myasnikov AL, Berns SA, Talyzin PA, Ershov FI. [Interferon gamma in the treatment of patients with moderate COVID-19]. Vopr Virusol. 2021 Mar 7;66(1):47-54. doi: 10.36233/0507-4088-24. Russian. PMID 33683065
- [Result] Myasnikov AL, Berns SA, Erhshov FI. Clinical application of interferon gamma in comprehensive therapy of patients with coronavirus infection. Rossiiskii meditsinskii zhurnal (Medical Journal of the Russian Federation, Russian Journal). 2020;26(6):394-401.